CLINICAL TRIAL: NCT00658307
Title: The Effects of Repetitive Transcranial Magnetic Stimulation in Healthy Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Z. J. Daskalakis, Chair, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 009/2008
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: repetitive transcranial magnetic stimulation; double-blind; sham-controlled; randomized
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- 2 (Experimental)
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- 3 (Sham Comparator)
  Interventions: Device: sham repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — 1 Hz
  The rTMS device is the "MagPro X100 Series" (produced by Magventure A/S, Farum, Denmark)
  Other Names: MagPro X100 Series
  Arms: 1
Device: repetitive transcranial magnetic stimulation (rTMS) — 20Hz
  The rTMS device is the "MagPro X100 Series" (produced by Magventure A/S, Farum, Denmark)
  Other Names: MagPro X100 Series
  Arms: 2
Device: sham repetitive transcranial magnetic stimulation (rTMS) — The rTMS device is the "MagPro X100 Series" (produced by Magventure A/S, Farum, Denmark)
  Other Names: MagPro X100 Series
  Arms: 3

SUMMARY:
It has been suggested that the therapeutic effects of repetitive transcranial magnetic stimulation (rTMS) are mediated through changes in cortical inhibition (CI). However, in healthy subjects the effects of rTMS on CI have been inconsistent. The aim of this study is to explore different rTMS - stimulus conditions neurophysiological and molecular mechanisms in the human motor cortex. Fifty-six healthy subjects will be randomized into three different treatment groups and receive 1 active or sham rTMS session (6000 rTMS pulses) at 90% of their motor threshold (MT). Cortical inhibition will be indexed pre and post treatment using short-interval intracortical inhibition (SICI), cortical silent period (CSP) and long-interval cortical inhibition (LICI).

Based on previous studies we hypothesize that:

* Hypothesis 1: rTMS will result in a greater CI (i.e., prolonged CSP, increased LICI but not SICI) compared to sham rTMS.
* Hypothesis 2: 20 Hz rTMS will result in a significantly greater CI compared to 1 Hz rTMS.
* Hypothesis 3: There will be distinctive transcription profiles associated with increases in CI from rTMS that can be detected with whole-genome microarray analysis of peripheral leukocytes.

DETAILED DESCRIPTION:
It has been demonstrated that several neurologic and psychiatry disorders are associated with dysfunctional cortical inhibitory mechanisms and alterations in neurotrophins (biological markers involved in neuronal survival and plasticity) and that rTMS therapeutic effects are associated with changes in cortical excitability. CI produced by rTMS can be demonstrated through SICI, CSP and LICI. However it remains unclear which rTMS parameters induce the best CI. Exploring different rTMS stimulus conditions versus sham condition effects in CI of human motor cortex can be the way to identify the best rTMS therapeutic parameters. Also, evaluating the molecular effects produced by rTMS treatment on serum blood levels can help identify the mechanisms through which rTMS exerts its therapeutic effects and ultimately clarify mechanisms through which treatment effects are mediated.

This experiment intends to demonstrate the best rTMS parameters to acquire higher CI. If our hypotheses are correct, these parameters will help to obtain higher therapeutic effects, and consequently, improvement of rTMS treatments.

ELIGIBILITY:
Inclusion Criteria:

* are voluntary and competent to consent
* between the ages of 18-65
* considered a healthy individual free of psychopathology based on the Personality Assessment Inventory
* right-handed determined by the TMS-screener and demographic form
* self-reported non-smoker
* do not have a self-reported concomitant major medical or neurologic illness
* women in childbearing years will be recruited only if they are on an effective means of birth control determined through completion of the TMS screener and demographic form.

Exclusion Criteria:

* demonstrate a failure to tolerate the procedure
* develop any significant adverse events (e.g., seizure or seizure-like activity)
* withdraw consent
* the principal investigator believes that for safety reasons it is in the best interest of the individual to be withdrawn

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Changes in CI produced by different frequency of stimulus and duration of treatments indicated by LICI, CSP and SICI | intermittent

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Daskalakis, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research